CLINICAL TRIAL: NCT02769845
Title: Stroke Avoidance for Children in REpublica Dominicana (SACRED): A Prospective Research Study to Reduce Stroke in Children With Sickle Cell Anemia
Brief Title: SACRED A Prospective Research Study to Reduce Stroke in Children With Sickle Cell Anemia
Acronym: SACRED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Hospital Infantil Dr. Robert Reid Cabral (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015-8767 SACRED
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longitudinal Portion (Experimental): All enrolled children will undergo yearly TCD examination. The goal of serial examination is to help define the natural history of cerebrovascular disease, specifically to determine the incidence of new conditional or abnormal velocities. The goal is to obtain a total of 3 TCD examinations per enrolled patient, regardless of treatment status.
  Interventions: Procedure: TCD examination
- Treatment Phase (Experimental): Those children with TCD velocities between 170-199 cm/sec will be eligible for protocol-directed hydroxyurea therapy. Most participants will initiate hydroxyurea treatment but those who are already on hydroxyurea and have conditional velocities will receive dose optimization. Participants will be followed until a common study termination date, defined as 3 years from the first treatment. Participants with abnormal TCD velocities ≥200 cm/sec will commence with transfusion therapy per current practice guidelines at the clinical site. Patients already on transfusion therapy identified to have conditional velocities will also be eligible for hydroxyurea and those with abnormal velocities may require re-calculation of transfusion dosing.
  Interventions: Drug: Hydroxyurea; Procedure: TCD examination

INTERVENTIONS:
Drug: Hydroxyurea — drug to be administered
  Arms: Treatment Phase
Procedure: TCD examination — TCD examinations on children with SCA between ages 3-15 years will be completed to evaluate their risk of stroke. All enrolled children will undergo yearly TCD examination. Participants with conditional TCD velocities on hydroxyurea therapy per study protocol will undergo TCD examinations every 6 months.

SUMMARY:
Prospective screening and treatment study for children with Sickle Cell Anemia and increased stroke risk living in the Dominican Republic.

DETAILED DESCRIPTION:
SACRED involves a three-part study design, as outlined below, to include (1) initial TCD evaluation phase; (2) longitudinal TCD evaluation; and (3) treatment if warranted.

1. The initial evaluation portion of SACRED will involve obtaining TCD examinations on children with SCA between ages 3-15 years, who are followed at Hospital Infantil Robert Reid Cabral in Santo Domingo to evaluate their risk of stroke. Up to 500 patients will be enrolled. All patients, including those who are already on hydroxyurea and transfusion therapy (whether for stroke or other clinical indications), will be included to obtain a one-year cross-sectional description of TCD velocities in this patient population. Patients who are already on therapy and identified to have elevated TCD velocities will be eligible for the treatment portion of SACRED as a conditional or elevated velocity would suggest that their present therapy was not optimized.
2. In the longitudinal portion of SACRED, all enrolled children will undergo yearly TCD examination. The goal of serial examination is to help define the natural history of cerebrovascular disease, specifically to determine the incidence of new conditional or abnormal velocities. The goal is to obtain a total of 3 TCD examinations per enrolled patient, regardless of treatment status.
3. In the treatment phase of SACRED, those children with TCD velocities between 170-199 cm/sec will be eligible for protocol-directed hydroxyurea therapy. Most participants will initiate hydroxyurea treatment but those who are already on hydroxyurea and have conditional velocities will receive dose optimization. Participants will be followed until a common study termination date, defined as 3 years from the first treatment. Participants with abnormal TCD velocities ≥200 cm/sec will commence with transfusion therapy per current practice guidelines at the clinical site. Patients already on transfusion therapy identified to have conditional velocities will also be eligible for hydroxyurea and those with abnormal velocities may require re-calculation of transfusion dosing.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric participants with severe forms of sickle cell anemia (HbSS or HbSβ° thalassemia)
* Age: between 3.0 and 15.0 years at the time of enrollment
* Parent or guardian willing and able to provide informed consent
* Ability to comply with study related treatments, evaluations, and follow-up

There are no exclusion criteria applicable to the TCD screening portion of SACRED.

For participants with conditional TCD velocities, the following criteria will disqualify them from the treatment phase of SACRED:

Exclusion Criteria:

* Known medical condition making participation ill-advised (e.g., acute or chronic infectious disease including HIV, known allergy to hydroxyurea therapy, or malignancy)
* Abnormal historical laboratory values (most recent pre-enrollment values):

  1. Anemia: Hemoglobin concentration < 6.0 gm/dL
  2. Reticulocytopenia: Absolute reticulocyte count < 100 x 10˄9/L with a hemoglobin concentration < 8.0 gm/dL
  3. Neutropenia: Absolute neutrophil count (ANC) < 1.0 x 10˄9/L
  4. Thrombocytopenia: Platelet count < 80 x10˄9 /L
  5. Known abnormal renal function (serum creatinine >2X upper limit for age AND ≥ 1.0 mg/dL)
* Pregnancy (for post-menarchal females only)

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Transcranial Doppler Ultrasound examinations | 0-24 months
  Serial TCD velocities will be measured yearly for participants not receiving hydroxyurea and every six months for participants receiving hydroxyurea during the trial. The outcome measure will be the highest TAMV obtained in the main intracranial arteries: middle cerebral artery (MCA), internal carotid artery (ICA), or internal carotid bifurcation (BIF). Subsequent TCD velocities will be compared to the baseline TCD values to describe the potential efficacy of hydroxyurea to reduce elevated TCD velocities.

SECONDARY OUTCOMES:
Hydroxyurea toxicities | 0-30 months
  This measure will be performed at least quarterly throughout the trial, and monthly during dose escalation by recording the CBC and Retic count.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Encargada del Servicio de Hematología-Oncología Hospital Infantil Dr. Robert Reid Cabral, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nieves RM, Latham T, Marte N, Berges M, Sanchez LM, Urcuyo G, Florencio C, Gonzalez C, Del Villar P, Chen S, Ramirez D, Reyes P, Marinez M, Matos E, Jeste ND, Stuber SE, Schultz WH, Lane AC, Mena R, Ware RE. Stroke prevention in Hispanic children with sickle cell anemia: the SACRED trial. Blood Adv. 2025 Apr 22;9(8):1791-1800. doi: 10.1182/bloodadvances.2024014327. PMID 39820633
- [Derived] Jeste ND, Sanchez LM, Urcuyo GS, Berges ME, Luden JP, Stuber SE, Latham TS, Mena R, Nieves RM, Ware RE. Stroke Avoidance for Children in REpublica Dominicana (SACRED): Protocol for a Prospective Study of Stroke Risk and Hydroxyurea Treatment in Sickle Cell Anemia. JMIR Res Protoc. 2017 Jun 2;6(6):e107. doi: 10.2196/resprot.7491. PMID 28576754